CLINICAL TRIAL: NCT05638659
Title: Elucidate the Mechanisms, Development and Effectiveness of Balance Control and Gait Strategy After Mild Traumatic Brain Injury: Develop Innovative Design of Computerized Dual-task Balance Module
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Li-Fong Lin, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202201026
Record Dates: First submitted 2022-10-13; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Twice a week for 8 weeks, total of 16 sessions course of computerized dual-task balance and home program.
  Interventions: Behavioral: Computerized dual-task balance and home program
- Control group (Active Comparator): Medical consultation and traditional balance training, and assessed after 8 weeks.
  Interventions: Behavioral: Medical consultation and traditional balance training

INTERVENTIONS:
Behavioral: Computerized dual-task balance and home program — Portable force plate with aluminum top plate for measuring ground reaction forces, moments and the center of pressure in biomechanics. Through software to collect data from the force plates, converts the trials into useful information and plots the results. The force plates and charge amplifiers are fully remote controlled by software thus making the system extremely flexible and easy to use.
  Arms: Experimental group
Behavioral: Medical consultation and traditional balance training — Participants were assigned to read the health education flier and were assessed directly.
  Arms: Control group

SUMMARY:
The purpose of this study is to innovatively design and develop computerized dual-task balance training modules and home modules, and conduct proactive clinical verification to focus on the effectiveness of balance control and gait stabilization strategies. It is expected that in addition to the development of the training module, a proactive study will be conducted at the same time. During the period from the fourth quarter of the first year to the second year, there will be 25 patients in the experimental group and 25 patients in the control group. A total of 50 patients will undergo preliminary efficacy analysis.

DETAILED DESCRIPTION:
After mild traumatic brain injury (mTBI), patients often complain of dizziness, balance disturbances, and gait instability. On average, dizziness accounts for about 23 to 81%, and dizziness symptoms persist from 1.2% 6 months after the injury. Between 32.5% in 5 years. In the past, in the process of neuron regeneration and repair after mild traumatic brain injury, it was found that vestibular function and biomarkers may be related to balance restoration and treatment. It is necessary to conduct further research to explain its potential mechanism and clinical significance. In addition, balance training after mTBI can accelerate dizziness recovery, balance control and gait stability, but the effect lasts for a limited time. The development of a dual-task balance training module can extend the recovery time, this project needs to be discussed in depth. This project mainly explores the influence of balance control and gait strategies after mTBI, linking vestibular function and biomarkers; innovative design and development of computerized dual-task balance training and home modules; combined with computerized dual-task balance training modules can accelerate the recovery of dizziness, balance control and gait stability after injury.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80 years old.
* Patients with mild traumatic brain injury: According to the American Congress of Rehabilitation Medicine, the loss of consciousness is less than 30 minutes, the coma index is 13-15, and the post-traumatic amnesia is less than 24 hours.
* Healthy patients: healthy subjects without any neurological, psychiatric, or severe musculoskeletal medical history.
* Regardless of gender.

Exclusion Criteria:

* Mild traumatic brain injury: moderate to severe brain injury, epilepsy, history of cardiovascular disease, lack of intelligence, neurodegenerative diseases, history of head trauma, systemic diseases, left-handedness, and use of psychotropic drugs.
* Healthy subjects: any neurological, psychiatric, severe musculoskeletal medical history.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Balance test | The end of intervention (assessments within one week)
  Berg Balance Scale (BBS), which rated performance from 0 (cannot perform) to 4(normal performance) on 14 different tasks, including ability to sit, stand, reach, lean over, turn and look over each shoulder, turn in a complete circle and step. The total possible score is 56, indicating excellent balance. A score of 0 to 20 indicates a high risk, 21 40 indicates a medium risk, and 41 56 indicates a low risk of falling. indicates a low risk of falling. Balance Error Scoring System (BESS) test Balance Error Scoring System (BESS) test
Balance of sensory-integration test | The end of intervention (assessments within one week)
  The balance of postural-stability test and the modified clinical test of sensory integration and balance (mCTSIB) were performed using the Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA).
Balance of postural-stability test | The end of intervention (assessments within one week)
  The balance of postural stability was tested according to 3 stability indices (overall stability, OA; anterior-to-posterior stability, AP; and medial-to-lateral stability, ML).
Modified clinical test of sensory integration and balance (mCTSIB) | The end of intervention (assessments within one week)
  The mCTSIB, which includes 4 sway indices, was conducted 4 sensory conditions: (1) eyes open whilst standing on a firm surface (EOFIS); (2) eyes closed whilst standing on a firm surface (ECFIS); (3) eyes open whilst standing on an unstable (foam) surface (EOFOS); and (4) eyes closed whilst standing on an unstable (foam) surface (ECFOS).
Gait analysis | The end of intervention (assessments within one week)
  The spatiotemporal gait parameters of asymmetry of the feet were measured with Physilog® system (Gait up Sàrl, Lausanne, Switzerland).
Vestibular function test - oculomotor system | The end of intervention (assessments within one week)
  Use smooth pursuit eye movements (SPEMs) to obtain baseline data. The examiner evaluates SPEMs by subjectively noting their accuracy in relation to a target that is being moved manually to nine directions. At the same time, the patient follows it with his or her eyes.

SECONDARY OUTCOMES:
Biomarker | The end of intervention (assessments within one week)
  Sera were assessed for for anti-bone marrow X kinase (anti-BMX, or cytoplasmic tyrosine-protein kinase) antibodies using using a commercial enzyme-linked immunosorbent assay (ELISA) kit with a range of 1.56 g/L according to the manufacturer's instructions. Results were determined by the optical density of each well, using the microplate reader Infinite 200 measured at 450 nm. A standard curve was made by reducing the data using the computer software Magellan capable of generating a four-parameter logistic (4-PL) curve-fit and calculating the sample concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan